CLINICAL TRIAL: NCT01124305
Title: A Prospective, Randomized Evaluation of Total Knee Arthroplasty Performed With Conventional and Customized Patient Instrumentation
Brief Title: Knee Arthroplasty Performed With Conventional and Customized Instrumentation
Acronym: CPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Responsible Party: Principal Investigator, Nancy Parks, Knee Project Director, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AORI2010-0101
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-11

CONDITIONS: Knee Arthritis
Keywords: Total Knee Arthroplasty; Instrumentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Instrumentation (Active Comparator): Control group: Cases performed with traditional surgical instruments
  Interventions: Device: Traditional Instrumentation
- Customized Patient Instrumentation (Experimental): Experimental group: Cases performed with custom instruments specifically made for each patient using pre-op CT scans.
  Interventions: Device: Customized Patient Instrumentation

INTERVENTIONS:
Device: Customized Patient Instrumentation — Custom cutting guides based on computed tomography (CT) images of the patient's leg are used to make the bone cuts and select the implant size.
  Arms: Customized Patient Instrumentation
Device: Traditional Instrumentation — Traditional surgical instruments will be used to make bone cuts and size the components in this control group.
  Arms: Traditional Instrumentation

SUMMARY:
The main purpose of this study is to determine whether the surgical time required for primary total knee arthroplasty is significantly less when performed with Customized Patient Instrumentation (CPI) than with conventional instrumentation. Each case will be recorded by video camera, in order to time the length of surgery and each surgical step. The number of surgical trays required for each case will be recorded. As an additional endpoint, the investigators will measure limb and component alignment on x-rays to determine if these two methods achieve equivalent alignment results. The thickness of bone cuts will be compared to the surgical plan and to each other.

The primary hypothesis is that the use of customized patient instrumentation will reduce the operative time required for total knee arthroplasty.

DETAILED DESCRIPTION:
Patient-specific instrumentation (PSI) has been developed for total knee arthroplasty (TKA) with several potential advantages over traditional instrumentation (TI). Shortened surgical time, fewer surgical instruments, and improved alignment are some of these proposed advantages. We sought to examine these assertions.

52 patients (26 per group) were enrolled in a prospective, randomized trial comparing CT-based PSI with TI. No difference was seen in average patient age (68 years) or BMI (31) between groups (p=0.84 and p=0.89), although there were more males in the PSI group (14 vs 7, p=0.002). A single surgeon and consistent staff performed the surgeries with the same knee prostheses, and all cases were videotaped to measure the length of surgery and each individual step. Any additional bone cuts, size changes, or ligament releases made to achieve correct alignment and balance were documented. The number of instrument trays opened for each case was recorded. Postoperative long alignment and lateral radiographs were taken to measure the coronal and sagittal plane component alignment and mechanical axis in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires unilateral primary total knee arthroplasty

Exclusion Criteria:

* Body mass index greater than 41
* Previous ipsilateral hip or ankle replacement
* Knee flexion contracture greater than 20 degrees

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Hamilton, MD, Principal Investigator — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States

REFERENCES:
- [Background] Lombardi AV Jr, Berend KR, Adams JB. Patient-specific approach in total knee arthroplasty. Orthopedics. 2008 Sep;31(9):927-30. doi: 10.3928/01477447-20080901-21. No abstract available. PMID 18814618
- [Background] Ng VY, DeClaire JH, Berend KR, Gulick BC, Lombardi AV Jr. Improved accuracy of alignment with patient-specific positioning guides compared with manual instrumentation in TKA. Clin Orthop Relat Res. 2012 Jan;470(1):99-107. doi: 10.1007/s11999-011-1996-6. PMID 21809150
- [Background] Howell SM, Kuznik K, Hull ML, Siston RA. Results of an initial experience with custom-fit positioning total knee arthroplasty in a series of 48 patients. Orthopedics. 2008 Sep;31(9):857-63. doi: 10.3928/01477447-20080901-15. PMID 18814593
- [Background] Bali K, Walker P, Bruce W. Custom-fit total knee arthroplasty: our initial experience in 32 knees. J Arthroplasty. 2012 Jun;27(6):1149-54. doi: 10.1016/j.arth.2011.12.006. Epub 2012 Jan 27. PMID 22285230
- [Background] Watters TS, Mather RC 3rd, Browne JA, Berend KR, Lombardi AV Jr, Bolognesi MP. Analysis of procedure-related costs and proposed benefits of using patient-specific approach in total knee arthroplasty. J Surg Orthop Adv. 2011 Summer;20(2):112-6. PMID 21838072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a suburban orthopaedic clinic setting between June 2010 and Sept 2011.
Pre-assignment Details: Patients were excluded if their medical insurance did not cover a leg CT scan or if there was any metal in their leg.
Period: Overall Study
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation
Started | 34 | 36
Completed | 26 | 26
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (12.1) | 69.2 (8.5) | 70.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 11 | 17 | 28
Region of Enrollment [Number; unit: participants]
  United States | 34 | 36 | 70

OUTCOME MEASURES:

1. Primary Outcome: Length of Surgery
Description: Time elapsed from skin incision to wound closure (in seconds)
Time Frame: 1 day
Population: per protocol
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation
Number analyzed (Participants) | 26 | 26
seconds | 3447.19 (297.68) | 3707.19 (348.26)

2. Secondary Outcome: Length of Each Surgical Step (in Seconds)
Description: surgical exposure, tibial alignment and resection, femoral distal cut, extension gap balancing, sizing the femur, 4 finishing femoral cuts, posterior releases, patellar resection, trial components, tibial tray preparation, cleanup/ prep for cement, cementing femur, cementing tibia, cementing patella, and closure
Time Frame: 1 day
Population: per protocol
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation
Number analyzed (Participants) | 26 | 26
seconds
  Exposure | 297.19 (54.87) | 318.38 (64.00)
  Tibial Alignment and Resection | 111.77 (37.67) | 129.73 (29.47)
  Femoral Distal Cut | 95.19 (19.5) | 170.46 (86.91)
  Extension Gap Balancing | 89.77 (73.88) | 77.88 (59.35)
  Sizing the Femur | 41.58 (11.70) | 21.46 (42.01)
  4 Finishing Femoral Cuts | 135.54 (35.67) | 186.96 (89.69)
  Posterior Releases | 225.42 (46.91) | 223.81 (51.68)
  Patellar Resection | 133.04 (27.51) | 136.31 (30.41)
  Trial Components | 247.92 (64.76) | 253.42 (78.78)
  Tibial Tray Preparation | 71.85 (24.20) | 67.54 (24.38)
  Cleanup/ Prepare for Cement | 206.46 (59.32) | 196.00 (53.16)
  Cementing Femur | 127.15 (22.86) | 141.65 (22.55)
  Cementing Tibia | 77.77 (16.99) | 83.62 (18.47)
  Cementing Patella | 102.65 (45.14) | 97.77 (22.98)
  Closure | 1221.62 (140.27) | 1246.69 (133.82)

3. Secondary Outcome: Number of Instrument Trays Required
Time Frame: 1 day
Population: per protocol
Measure: Mean (Standard Deviation); unit: number of trays
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation
Number analyzed (Participants) | 26 | 26
number of trays | 7.3 (0.69) | 2.5 (1.14)

4. Secondary Outcome: Limb Alignment (Mechanical Axis)
Description: Alignment is measured on 4 month postoperative radiograph in degrees. The goal is a mechanical axis between and femur and tibia of 0 degrees. Varus alignment ("bow-legged") is shown as a negative number in degrees away from 0. Valgus alignment ("Knock-kneed") is expressed as a positive number in degrees away from 0.
Time Frame: 4 months
Population: All participants were x-rayed postoperatively to measure the mechanical axis of the leg in degrees.
Measure: Mean (Full Range); unit: degrees varus(-) or valgus(+)
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation
Number analyzed (Participants) | 26 | 26
degrees varus(-) or valgus(+) | 0.7 [-5.9 to 7.6] | 0.3 [-6.8 to 6.4]

ADVERSE EVENTS:
Time Frame: 4 months
Description: This is a study of surgical instruments, therefore the focus would be on adverse events occurring during surgery. All patients were followed for 4 months, so we also able to capture adverse events in the short-term postoperative period.
Arm/Group | Traditional Instrumentation | Customized Patient Instrumentation
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 1/26 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Instrumentation (N=26) | Customized Patient Instrumentation (N=26)
Knee stiff (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Manipulation under anesthesia for limited range of motion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No